CLINICAL TRIAL: NCT04676360
Title: A Multicenter Phase 2 Study of Belantamab Mafodotin in Relapsed or Refractory Plasmablastic Lymphoma and ALK+ Large B-cell Lymphoma
Brief Title: Belantamab Mafodotin In Plasmablastic Lymphoma & ALK+ Large B-Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed given lack of efficacy and plans to publish this negative study.
Sponsor: Jacob Soumerai, MD (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Jacob Soumerai, MD, Sponsor Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-404
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Relapsed Plasmablastic Lymphoma; Refractory Plasmablastic Lymphoma; Anaplastic Lymphoma Kinase Positive Large B-Cell Lymphoma
Keywords: Relapsed Plasmablastic Lymphom; Refractory Plasmablastic Lymphoma; Anaplastic Lymphoma Kinase Positive Large B-Cell Lymphoma
MeSH Terms: conditions — Plasmablastic Lymphoma | interventions — belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- (BELANTAMAB MAFODOTIN (Experimental): * Belantamab mafodotin will be administered intravenously on day 1 of a 21-day cycle.
  * Treatment is intended to be administered on an outpatient basis.
  Interventions: Drug: Belantamab Mafodotin

INTERVENTIONS:
Drug: Belantamab Mafodotin — Belantamab mafodotin will be administered intravenously at calculated dose on day 1 of each 21-day cycle.
  Other Names: Blenrep

SUMMARY:
In this research study is looking to see how safe and effective belantamab mafodotin is in relapsed or refractory plasmablastic lymphoma or ALK+ large B-cell lymphoma.

* This research study involves the study drug belantamab mafodotin.
* Belantamab mafodotin is an antibody-drug conjugate (ADC), which is the combination of an antibody (a protein that binds to cells) and a drug. It works by using the antibody portion to enter into the lymphoma cells, and then releasing the drug portion to kill the lymphoma cells.

DETAILED DESCRIPTION:
This is a multicenter phase 2 study of belantamab mafodotin on participants with plasmablastic lymphoma and ALK+ large B-cell lymphoma.The research study procedures include screening for eligibility, and study treatment, including evaluations and follow up visits.

* This research study involves the study drug belantamab mafodotin.
* Participants may receive the study treatment until progression or intolerance, and will be followed up to 2 years.
* It is expected that about 25 people will take part in this research study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved belantamab mafodotin as a treatment for any disease. This study drug is investigational, and it is not known whether participants will benefit from taking belantamab mafodotin.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have relapsed or refractory plasmablastic lymphoma or ALK+ large Bcell lymphoma by WHO criteria.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter [LDi] to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥15 mm in LDi for nodal disease or ≥10 mm in LDi for extranodal lesions.
* Participants must have received prior systemic lymphoma therapy.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of belantamab mafodotin in participants <18 years of age, children are excluded from this study.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Participants must have adequate marrow function as defined below (unless abnormalities are considered related to marrow and/or splenic involvement by lymphoma):

  * absolute neutrophil count ≥1,000/mcL
  * platelets ≥50,000/mcL
  * hemoglobin ≥ 8.0 g/dL
* Participants must have adequate organ function as defined below:

  * total bilirubin ≤ 1.5 X institutional upper limit of normal (ULN); (Isolated bilirubin ≥1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN
  * Spot urine (albumin/creatinine) <500 mg/g (56 mg/mmol) OR
  * Urine Dipstick Negative/trace (if ≥1+ only eligible if confirmed ≤ 500 mg/g (56 mg/mmol) by albumin/creatinine ratio (spot urine from first void)
  * Glomerular filtration rate (eGFR)≥30 mL/min/1.73 m2 (MDRD Formula).
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Belantamab mafodotin is potentially teratogenic. A female participant is eligible to participate if she is not pregnant or breastfeeding. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 4 months after the last dose of study intervention. Women must also agree not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Nonchildbearing potential is defined as follows (by other than medical reasons):

  * ≥45 years of age and has not had menses for >1 year
  * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.
* Women of childbearing potential must have a negative highly sensitive serum pregnancy test, and agree to repeat highly sensitive serum pregnancy testing within 72 hours before the first dose of study intervention (if screening pregnancy test was not within 72 hours of dosing).
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of administration. Men must also agree not to donate sperm during this period. Men may agree to remain abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) OR agree to use a male condom, even if they have undergone a successful vasectomy and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year when having sexual intercourse with a WOCBP (including pregnant females).
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial at the discretion of the overall PI.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants must not have current corneal epithelial disease except mild changes in corneal epithelium.
* Participant must not have current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable non cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia. At the discretion of the overall PI, participants with residual toxicities > Grade 1 may be considered eligible if in the opinion of the overall PI the residual toxicity is not likely to interfere with the safety or efficacy assessment of the investigational regimen.
* Participants who are receiving any other investigational agents.
* Participants must not have central nervous system involvement by lymphoma, as belantamab mafodotin is not known to penetrate the CNS.
* Participant must not use contact lenses while participating in this study.
* Participant must not be simultaneously enrolled in any interventional clinical trial.
* Participant must not have used an investigational drug or approved systemic lymphoma therapy within 14 days or five half-lives, whichever is shorter, preceding the first dose of study drug. Steroids are permitted.
* Participant must not have had major surgery within 4 weeks of initiating study treatment.
* Participant must not have any evidence of active mucosal or internal bleeding.
* Participants must not have known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to belantamab mafodotin or drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.
* Participants must not have an uncontrolled intercurrent illness.
* Participant must not have an uncontrolled active infection.
* Participant must not have evidence of cardiovascular risk including any of the following:

  * Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block.
  * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting/bypass grafting within three (3) months of Screening.
  * Class III or IV heart failure as defined by the New York Heart Association functional classification system [NYHA, 1994].
  * Participant must not have uncontrolled hypertension defined as persistent systolic BP >160 mmHg or diastolic BP >100 mmHg.
* Participant must not have psychiatric illness/social situations that would limit compliance with study requirements. Participants must not have any serious and/or pre-existing medical or other condition (including lab abnormalities) that could interfere with participant's safety in the opinion of the investigator.
* Women who are pregnant or lactating are excluded from this study because belantamab mafodotin can cause embryo-fetal harm when administered to a pregnant woman. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with belantamab mafodotin, breastfeeding should be discontinued if the mother is treated with belantamab mafodotin.
* Participant must not have presence of hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb) at screening or within 3 months prior to first dose of study treatment. Patients with presence of HBsAg, but demonstrate both HBSag and HBV PCR negativity will be eligible for the study. Participant must not have positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment. Note: Participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained. Note: Hepatitis RNA testing is optional and participants with negative Hepatitis C antibody test are not required to also undergo Hepatitis C RNA testing.
* Participant must not have uncontrolled HIV infection. HIV-infected patients on effective anti-retroviral therapy are eligible if they (1) have an undetectable viral load within the prior 6 months, or (2) have a detectable viral load with an absolute CD4 count of 200 cells per microliter or higher.
* Participant must not have invasive malignancies other than disease under study, unless the second malignancy has been medically stable for at least 2 years and, in the opinion of the principal investigators, will not affect the evaluation of the effects of clinical trial treatments on the currently targeted malignancy. Participants with adequately treated basal, squamous cell carcinoma or non-melanomatous skin cancer, carcinoma in situ of the cervix, superficial bladder cancer not treated with intravesical chemotherapy or BCG within 6 months, localized prostate cancer and PSA <1.0 mg/dL on 2 consecutive measurements at least 3 months apart with the most recent one being within 4 weeks of study entry, may be enrolled without a 2-year restriction.
* Participant must not have had plasmapheresis within 7 days prior to first dose of study treatment
* Participant must not have received prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Screening; after 2 months; after 4 months, after 6 months; then every 6 months on therapy up 2 years
  An objective response rate (ORR, PR or better) of at least 30% will be considered promising whereas an ORR of 10% or less will be considered non-promising. The responses will classified per the 2014 Lugano criteria. The frequency of complete response will be tabulated and summarized descriptively.

SECONDARY OUTCOMES:
Complete Response Rate | Screening; after 2 months; after 4 months, after 6 months; then every 6 months on therapy up 2 years
  Patients will have their response classified per the 2014 Lugano criteria. The frequency of complete response will be tabulated and summarized descriptively.
Progression Free Survival | Participants will be followed for 2 years after removal from protocol therapy or until death, whichever occurs first up to 4 years
  Median Progression-free survival will be summarized using Kaplan-Meier method with time of registration as time origin. Participants will be followed for 2 years after removal from protocol therapy or until death, whichever occurs first. Participants will be censored at the date of their last evaluation.
Overall Survival | Participants will be followed for 2 years after removal from protocol therapy or until death, whichever occurs first up to 4 years
  Overall survival will be summarized using Kaplan-Meier method with time of registration as time origin. Participants will be followed for 2 years after removal from protocol therapy or until death, whichever occurs first. Participants will be censored at the date of their last evaluation.
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v5.0 | start of study treatment until at least 70 days following End of Treatment up to 2 years
  Patients will have their toxicities graded and reported at every visit according to criteria listed in CTAE ver. 5.0. The nature, frequency, severity, and timing of adverse events will be tabulated and summarized descriptive

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Soumerai, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation